CLINICAL TRIAL: NCT07405411
Title: The Prevalence, Causes, and Prevention Strategies of Medical Malpractice in Psychiatric Clinics: A Descriptive and Correlational Study
Brief Title: The Prevalence, Causes, and Prevention Strategies of Medical Malpractice in Psychiatric Clinics
Status: Completed | Type: Observational
Sponsor: Abant Izzet Baysal University (Other)
Responsible Party: Principal Investigator, Melisa BULUT, Research Assistant PhD, Abant Izzet Baysal University
Other Study IDs: AIBU-PSK-MB-03
Record Dates: First submitted 2025-09-18; First posted 2026-02-12 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Psychiatric Hospitalization; Patient Safety
Keywords: malpractice; medical practice errors; psychiatry; patient safety

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Malpractice in psychiatry is the failure of mental health professionals to meet accepted standards of care, resulting in harm to patients. While considered less risky than other specialties, the nature of psychiatry presents unique challenges and legal risks.

This descriptive and cross-sectional study investigated the frequency, influencing factors, and attitudes regarding medical malpractice among psychiatrists, residents, and nurses in psychiatric clinics in Turkey. Data was collected online via snowball sampling.

DETAILED DESCRIPTION:
This is a descriptive and cross-sectional study. Psychiatric professionals (psychiatrists, physician assistants, and clinical nurses) who had experience with malpractice in psychiatry and volunteered to share this experience were included in the study. Due to the sensitivity of the topic and the difficulty of accessing the sample, a snowball sampling method was used.

Participation Criteria:

Inclusion Criteria: Working in an inpatient psychiatric ward in Türkiye, having at least one year of experience in a psychiatric clinic, and agreeing to participate voluntarily.

Exclusion Criteria: Working in a child and adolescent psychiatry clinic.

Data Collection Tools:

Two forms developed by the researchers and validated for content validity were used:

Survey Form: Designed to assess participants' knowledge, attitudes, and behaviors on the subject. It consists of 22 questions. Validity: No items were removed because the "Content Validity Index (CVI), calculated using the Davis Technique and based on opinions from six experts, exceeded 0.80. Some items were revised based on expert suggestions. Reliability: Data were collected online to prevent participants from answering questions that measured knowledge by referring to definitional questions. Sensitivity: To overcome participant hesitancy, the questions were designed to ask whether they had witnessed a mistake, rather than who made the mistake.

Personal Information Form: This is a nine-question form designed to measure participants' individual characteristics, such as age, gender, occupation, and years of experience.

Data Collection Process: Data collection forms were sent online to participants who agreed to participate in the study and met the criteria.

ELIGIBILITY:
Inclusion Criteria:

* Working as a psychiatrist, assistant physician, or clinical nurse in any inpatient psychiatric service in Turkey,
* Having at least one year of experience in a psychiatric clinic
* Volunteering to participate in the study.

Exclusion Criteria:

* Working in a child and adolescent psychiatry clinic

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study recruited 180 participants (n=180), including psychiatrists, resident physicians continuing their psychiatric training, nurses, and psychiatric nurses working in psychiatric clinics in Turkey.
Sampling Method: Non-Probability Sample
Enrollment: 180 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2023-12-17 (Actual); Study Completion 2023-12-17 (Actual)

PRIMARY OUTCOMES:
malpractice frequency | Baseline
  The frequency of encountering malpractice cases among professionals working in psychiatric clinics

SECONDARY OUTCOMES:
causes of malpractice | Baseline
  Perceptions of professionals working in psychiatric clinics about the causes of malpractice cases
prevention strategies of medical malpractice | Baseline
  Perceptions of professionals working in psychiatric clinics about the prevention strategies of medical malpractice

CONTACTS AND LOCATIONS:
Overall Officials: Melisa Bulut, RN, PhD, Principal Investigator — Bolu Abant İzzet Baysal University
Locations (1):
- Faculty of Health Sciences, Bolu, Bolu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
May be made available upon request for appropriate data.Otherwise, the data will not be shared in the publication.

REFERENCES:
- [Background] Appelbaum PS. Malpractice claims in psychiatry: approaches to reducing risk. World Psychiatry. 2021 Oct;20(3):438-439. doi: 10.1002/wps.20907. No abstract available. PMID 34505366
- [Background] Dhadphale MR. Psychiatrist facing litigation. Indian J Psychiatry. 2019;61(4):405-408. doi: 10.4103/psychiatry.IndianJPsychiatry_316_17. PMID 31391646
- [Background] Aaron DG, Robertson CT, King LP, Sage WM. A New Legal Standard for Medical Malpractice. JAMA. 2025 Feb 26. doi: 10.1001/jama.2025.0097. Online ahead of print. PMID 40009364
- [Background] Frierson RL, Joshi KG. Malpractice Law and Psychiatry: An Overview. Focus (Am Psychiatr Publ). 2019 Oct;17(4):332-336. doi: 10.1176/appi.focus.20190017. Epub 2019 Nov 6. PMID 32047377
- [Background] Reuveni I, Pelov I, Reuveni H, Bonne O, Canetti L. Cross-sectional survey on defensive practices and defensive behaviours among Israeli psychiatrists. BMJ Open. 2017 Mar 20;7(3):e014153. doi: 10.1136/bmjopen-2016-014153. PMID 28320795